CLINICAL TRIAL: NCT00084591
Title: Phase I Study of Preoperative Intensity Modulated Radiation Therapy (IMRT) With Incorporated Boost and Oral Capecitabine in Locally Advanced Rectal Cancer
Brief Title: Intensity-Modulated Radiation Therapy With Incorporated Boost and Capecitabine Before Surgery in Treating Patients With Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000365462; P30CA006927 (NIH); FCCC-03606
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2010-02-12 (Estimated); Status verified 2010-02

CONDITIONS: Colorectal Cancer
Keywords: stage II rectal cancer; stage III rectal cancer; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: capecitabine
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Intensity-modulated radiation therapy (radiation directed at the tumor more precisely than in standard radiation therapy) with incorporated boost (an increase in the amount of radiation given during treatment) may cause less damage to normal tissue. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving radiation therapy together with chemotherapy before surgery may shrink the tumor so it can be removed.

PURPOSE: This phase I trial is studying the side effects and best dose of neoadjuvant intensity-modulated radiation therapy with incorporated boost when given together with capecitabine in treating patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of neoadjuvant boost intensity-modulated radiotherapy when combined with capecitabine before surgery in patients with locally advanced rectal cancer.

Secondary

* Determine the pathologic tumor response in patients treated with this regimen.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a dose-escalation study of boost intensity-modulated radiotherapy (IMRT).

Patients undergo neoadjuvant IMRT with incorporated boost once daily 5 days a week for 5 weeks. Beginning on the first day of radiotherapy, patients receive oral capecitabine twice daily 7 days a week for 5 weeks. Patients undergo surgical resection 4-8 weeks after completion of chemoradiotherapy.

Cohorts of 3-6 patients undergo escalating doses of boost IMRT until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 3 of 6 patients experience dose-limiting toxicity.

Quality of life is assessed at baseline, at week 5 of chemoradiotherapy, before surgery, and then at 1, 3, and 12 months after surgery.

Patients are followed at 1, 3, and 12 months after surgery.

PROJECTED ACCRUAL: Approximately 3-15 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary adenocarcinoma of the rectum

  * Distal border of the tumor within 12 cm of the anal verge by proctoscopic exam
  * Clinical stage T3-4, N1-2 (stage II or III) disease by 2 of the following tests:

    * Physical exam
    * Transrectal ultrasound
    * Pelvic CT scan
    * Pelvic MRI
* No clinical evidence of metastatic disease

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* No known, uncontrolled coagulopathy

Hepatic

* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* SGOT and SGPT ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal

* Creatinine ≤ 1.5 times normal
* Creatinine clearance > 50 mL/min

Cardiovascular

* No clinically significant cardiac disease
* No congestive heart failure
* No symptomatic coronary artery disease
* No poorly controlled cardiac arrhythmias
* No myocardial infarction within the past year

Gastrointestinal

* No active inflammatory bowel disease
* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome

Other

* No other prior or concurrent malignancy except inactive, non-invasive carcinoma of the cervix or non-melanoma skin cancer
* No concurrent serious, uncontrolled infection(s)
* No prior unanticipated severe reaction to fluoropyrimidine therapy
* No known sensitivity to fluorouracil
* No prior uncontrolled seizures
* No CNS disorders that would preclude study participation
* No other medical or psychiatric condition that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for rectal cancer

Chemotherapy

* No prior chemotherapy for rectal cancer

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy for rectal cancer
* No prior pelvic radiotherapy

Surgery

* More than 4 weeks since prior major surgery and recovered
* No prior surgery for rectal cancer

Other

* More than 4 weeks since prior participation in another investigational drug study
* No concurrent celecoxib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-12; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Acute toxicity by CTCAE at 6 weeks following study completion

SECONDARY OUTCOMES:
Quality of life as assessed by Quality of Life Questionnaire Core 30 Items (QLQ-C30) before and after radiotherapy and then every 6 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gary Freedman, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States